CLINICAL TRIAL: NCT00122707
Title: Randomized Controlled Trial of Mechanical and Infectious Complications of Central Versus Peripheral Venous Catheters in ICU Patients
Brief Title: Comparison of Central and Peripheral Venous Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LMR1
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2006-03-22 (Estimated); Status verified 2005-06

CONDITIONS: Respiratory Insufficiency; Shock; Coma
Keywords: catheter-related infection; mechanical complications of catheters
MeSH Terms: conditions — Respiratory Insufficiency; Shock; Coma; Catheter-Related Infections | interventions — Catheters

INTERVENTIONS:
Device: catheters

SUMMARY:
The purpose of this study is to compare the mechanical and infectious complications of peripheral versus central venous catheters in critically ill patients. Group allocation will be performed by randomization.

DETAILED DESCRIPTION:
Critically ill patients require intravenous administration of fluids and drugs. This can be achieved via peripheral or central catheters. Each device is associated with both mechanical and infectious complications. Complications associated with central lines are judged to be more severe. Some patients actually require the insertion of a central line due to the venous toxicity of the drugs or to the necessity of making sure that the infusion is regularly administered (example: high dose catecholamine infusion). Some physicians believe that most Intensive Care Unit (ICU) patients should have a central venous line inserted, whereas others feel that some patients may receive active drugs via a peripheral line in selected instances. No study prospectively compared the feasibility, merits and complications of the two possibilities (i.e., central or peripheral venous line). This study includes patients that can receive either a central or a peripheral line (see inclusion criteria): mainly patients receiving large amounts of fluid, moderate doses of catecholamines or of drugs that may cause venous injury. Patients are randomized to receive either a peripheral or a central venous catheter. Endpoints are the rate of mechanical complications (difficulty in inserting the line, need for repeat insertion attempts, occurrence of arterial puncture, occurrence of pneumothorax) and of infectious complications (local catheter infection or catheter-related bloodstream infection).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring low to moderate doses of continuous catecholamine administration in the ICU
* Patients with 2 failed attempts at inserting a peripheral line
* Patients who require daily change of lines

Exclusion Criteria:

* Patients aged less than 18 years
* Pregnancy
* Absolute necessity of central venous access (refractory shock/high dose catecholamine infusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-04; Study Completion 2005-10

PRIMARY OUTCOMES:
failure to insert line
mechanical complications of intravenous line insertion
infectious complications of intravenous lines

SECONDARY OUTCOMES:
number of cross-overs (due to impossibility of inserting/maintaining a peripheral line)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de Réanimation, Hopital Louis Mourier, Colombes, France

REFERENCES:
- [Background] Timsit JF. [Updating of the 12th consensus conference of the Societe de Reanimation de langue francaise (SRLF): catheter related infections in the intensive care unit]. Ann Fr Anesth Reanim. 2005 Mar;24(3):315-22. doi: 10.1016/j.annfar.2004.12.022. French. PMID 15792575
- [Background] Polderman KH, Girbes AJ. Central venous catheter use. Part 1: mechanical complications. Intensive Care Med. 2002 Jan;28(1):1-17. doi: 10.1007/s00134-001-1154-9. Epub 2001 Dec 4. PMID 11818994
- [Background] Polderman KH, Girbes AR. Central venous catheter use. Part 2: infectious complications. Intensive Care Med. 2002 Jan;28(1):18-28. doi: 10.1007/s00134-001-1156-7. Epub 2001 Nov 29. PMID 11818995
- [Derived] Ricard JD, Salomon L, Boyer A, Thiery G, Meybeck A, Roy C, Pasquet B, Le Miere E, Dreyfuss D. Central or peripheral catheters for initial venous access of ICU patients: a randomized controlled trial. Crit Care Med. 2013 Sep;41(9):2108-15. doi: 10.1097/CCM.0b013e31828a42c5. PMID 23782969